CLINICAL TRIAL: NCT06651736
Title: Optimizing Low Vision Rehabilitation in Emotionally Distressed Patients With Inherited Retinal Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, K. Thiran Jayasundera, Professor of Ophthalmology and Visual Sciences and Associate Chair, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00246479; 1R01EY035016-01A1 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Inherited Retinal Diseases
Keywords: Low Vision Rehabilitation; Emotional Regulation Therapy; Vision-related anxiety

STUDY DESIGN:
Intervention Model Description: Participants with IRD will be recruited and will be allocated into one of three study arms, depending on self-reported anxiety. Participants (N ~ 60) without vision-related anxiety will be designated to Arm 1 and receive LVR. Participants (N ~ 120) with vision-related anxiety will be randomly assigned to either Arm 2 or 3, in which participants will receive LVR with adjunctive ERT.
Who Masked: Care Provider
Masking Description: The 6 and 12-month post-LVR assessments will be administered by a study team member that is masked to Arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Low Vision Rehabilitation LVR (Active Comparator): Participants (N ~ 60) without vision-related anxiety will be designated to Arm 1 and receive LVR. This group is intended to be a comparison for the higher vision-related anxiety groups. For this reason, these patients may be placed on a waitlist (meaning participants low-vision rehabilitation may be delayed), until the study team can match with someone in one of the other groups.
  Interventions: Behavioral: Low Vision Rehabilitation (LVR)
- Arm 2 - ERT (after randomization) and then concurrent with LVR (Experimental): Participants with vision-related anxiety (must meet this per protocol by self-reports) randomized to this arm will receive immediate ERT. The LVR therapy will start approximately during 4-6 sessions of ERT.
  Interventions: Behavioral: Low Vision Rehabilitation (LVR); Behavioral: Emotion Regulation Therapy (ERT)
- Arm 3- LVR with delayed ERT (Experimental): Participants with vision-related anxiety (must meet this per protocol by self-reports) randomized to this arm will receive LVR with delayed ERT.
  Interventions: Behavioral: Low Vision Rehabilitation (LVR); Behavioral: Emotion Regulation Therapy (ERT)

INTERVENTIONS:
Behavioral: Low Vision Rehabilitation (LVR) — The initial session will be with an LVR specialist that will recommend vision-enhancing devices and techniques to improve participant's vision and mobility functionality depending on needs. The devices will be given at no cost and include, but are not limited to: magnifiers that participants can hold or wear, glasses attachments that help filter out light to see better, or items that help with glare or seeing color. This session will be followed by at least one session with an occupational therapist, that will train participants to use the devices (take home and use) and recommend/teach ways to achieve functional goals.
  Most participants will be asked to attend 2-4 visits, but additional visits may be needed depending on needs and progress toward functional goals. Additional visits if orientation and mobility training is also recommended. Participants will be asked to share experiences approximately 1-week after all visits.
Behavioral: Emotion Regulation Therapy (ERT) — There will be ten 1-hour weekly sessions of specialized psychotherapy with an ERT-trained therapist. These are typically done virtually but may be able to provide in-person sessions to those where this is needed. At the beginning of each session, the therapist will give participant's several questionnaires to learn about participant's experience with ERT. Questionnaires will also be completed after all sessions are completed.
  Arms: Arm 2 - ERT (after randomization) and then concurrent with LVR; Arm 3- LVR with delayed ERT

SUMMARY:
The purpose of this study is to understand if combining Low Vision Rehabilitation (LVR) with Emotional Regulation Therapy (ERT) can help people with inherited retinal diseases (IRDs) that experience emotional distress related to participants' vision loss.

The study team hypothesize that treatment with LVR will produce measurable functional gains and that these effects will be enhanced by ERT-linked improvement among the subgroup of IRD patients with elevated vision-related anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with vision impairment with IRD etiology
* Must have had a clinical exam with an IRD specialist within the three months of assignment to Arm
* Have had a Goldmann visual field that was tested with III-4e isopter within the last year
* Have a disability greater than zero theta in any of the domains of Michigan Retinal Dystrophy Questionnaire (MRDQ)
* Have an indication from the IRD specialist that the ocular condition will not deteriorate over the next 1- year
* Able to participate in 10 weeks of ERT sessions while being physically located in Michigan (these will take place in the first 10 months of the study)

Exclusion Criteria:

* Having other ocular comorbidities including those associated with an IRD such as control of cystoid macular edema (CME)
* Functional needs regarding low vision (i.e. activities of daily living) have been adequately addressed per a study low vision specialist
* Current mental health therapy
* The participant must not have an elevated suicidal intention (SI) or suicide risk based on Patient Health Questionnaire (PHQ-9) further information collected at screening (If suicidal intentions are identified, the study staff will complete the suicide protocol (per protocol)
* If the participant is using medication for mental health or psychiatry concerns, participants must be on a stable dose of the medication (1-month of taking), otherwise will be excluded
* Inability to complete study task requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2028-11-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Determine if LVR improves vision-related disabilities and distress measures by the Michigan Vision-related Anxiety Questionnaire (MVAQ) | Baseline to 6 month
  The Michigan Vision-related Anxiety Questionnaire is a 14 -item questionnaire designed to assess anxiety/distress related to vision impairments. Responses can range between: Never, Sometimes, Frequently, Always, N/A for Non-Vision Reasons. The questionnaire provides 2 scores (one for anxiety about rod function and one for anxiety about cone function). Both of those scores fall between -3 and 3 (an increasing score indicates higher levels of anxiety).
Determine if LVR improves vision-related disabilities and distress measures by the Michigan Retinal Degeneration Questionnaire (MRDQ) | Baseline to 6 month
  The Michigan Retinal Degeneration Questionnaire is a 59-item questionnaire aimed to assess vision-related functional impairment. Responses can range between: None, A little difficulty, Moderate difficulty, Extreme difficulty, My vision is too poor to do this, N/A for non-vision reasons. The questionnaire provides 7 scores (for 7 different domains of vision) and also range from -3 to 3 (0 is centered at the mean trait level of the population and extreme values for theta (i.e., -3, +3) are indicative of low or high visual dysfunction based on item responses).
Determine if LVR measures are different between low-distress and high-distress groups accessed at month-6 by MVAQ | Baseline, 6 months
  Comparison between low-distress arm and high-distress arm prior to ERT treatment at month-6. The Michigan Vision-related Anxiety Questionnaire is a 14 -item questionnaire designed to assess anxiety/distress related to vision impairments. The Michigan Vision-related Anxiety Questionnaire is a 14 -item questionnaire designed to assess anxiety/distress related to vision impairments. Responses can range between: Never, Sometimes, Frequently, Always, N/A for Non-Vision Reasons. The questionnaire provides 2 scores (one for anxiety about rod function and one for anxiety about cone function). Both of those scores fall between -3 and 3 (an increasing score indicates higher levels of anxiety).
Determine if LVR measures are different between low-distress and high-distress groups accessed at month-6 by MRDQ | Baseline, 6 months
  Comparison between low-distress arm and high-distress arm prior to ERT treatment at month-6.
  The Michigan Retinal Degeneration Questionnaire is a 59-item questionnaire aimed to assess vision-related functional impairment. Responses can range between: None, A little difficulty, Moderate difficulty, Extreme difficulty, My vision is too poor to do this, N/A for non-vision reasons. The questionnaire provides 7 scores (for 7 different domains of vision) and also range from -3 to 3 (0 is centered at the mean trait level of the population and extreme values for theta (i.e., -3, +3) are indicative of low or high visual dysfunction based on item responses).
Determine if adjunctive ERT treatment in the high-distress arms improves vision-related disabilities and vision-related distress measures greater than LVR alone measured by MVAQ | Baseline, 6 months
  The Michigan Vision-related Anxiety Questionnaire is a 14 -item questionnaire designed to assess anxiety/distress related to vision impairments. Responses can range between: Never, Sometimes, Frequently, Always, N/A for Non-Vision Reasons. The questionnaire provides 2 scores (one for anxiety about rod function and one for anxiety about cone function). Both of those scores fall between -3 and 3 (an increasing score indicates higher levels of anxiety).
Determine if adjunctive ERT treatment in the high-distress arms improves vision-related disabilities and vision-related distress measures greater than LVR alone measured by the MRDQ | Baseline, 6 months
  The Michigan Retinal Degeneration Questionnaire is a 59-item questionnaire aimed to assess vision-related functional impairment. Responses can range between: None, A little difficulty, Moderate difficulty, Extreme difficulty, My vision is too poor to do this, N/A for non-vision reasons. The questionnaire provides 7 scores (for 7 different domains of vision) and also range from -3 to 3 (0 is centered at the mean trait level of the population and extreme values for theta (i.e., -3, +3) are indicative of low or high visual dysfunction based on item responses).

SECONDARY OUTCOMES:
Determine if LVR improves vision-related disabilities and distress measures by the Short Form Survey (SF-36) | Baseline to 6 month
  The survey has 36-items in which participants select responses. It measures and produces scores (0-100) for 8 domains (Physical functioning, Role limitations due to physical health, Bodily pain, General health perceptions, Vitality (energy/fatigue), Social functioning, Role limitations due to emotional problems, Mental health (emotional well-being) Scores presented on a 0-100 scale, with scores above 50 generally indicating better-than-average health-related quality of life, and scores below 50 suggesting below-average health.
Determine if adjunctive ERT treatment improves LVR treatment adherence greater than LVR alone measured by the Psychosocial Impact of Assistive Devices Scale (PIADS) | 6 months
  The Psychosocial Impact of Assistive Devices (PIADS) is a 26-item self-reported questionnaire designed to assess the effects of an assistive device on functional independence, well-being and quality of life.
  The PIADS Uses a 7-point scale for each item, ranging from -3 to +3. A score of -3 indicates the maximum negative impact, a score of 0 indicates no impact or neutral effect, and a score of +3 indicates the maximum positive impact of devices.
Determine if adjunctive ERT treatment improves overall emotional distress greater than LVR alone measured by the Patient Health Questionnaire (PHQ-9) | 6 months
  The Patient Health Questionnaire is a 9-item questionnaire designed to assess depression symptoms. Participants answer questions from Not at all (0) -Nearly every day (3). The score ranges from 0 to 27, the higher scores mean more serious depression.
Determine if adjunctive ERT treatment improves overall emotional distress greater than LVR alone measured by the Perceived Stress Scale (PSS) | 6 months
  The Perceived Stress Scale is a 10-item questionnaire aimed to assess participants perceived stress. Items are scored from never (0) - very often (4). Scores rage from 0-40 with higher scores indicating higher stress.
Determine if adjunctive ERT treatment improves LVR treatment adherence greater than LVR alone measured by the Daughty Device Compliance Questionnaire (DDCQ) | 6 months
  The Daughty Device Compliance Questionnaire (DDCQ) is a 5-item self-reported questionnaire designed to evaluate the adherence to and effectiveness of medical devices in daily use. It assesses factors such as user satisfaction, ease of use, and the impact on health outcomes. Completed for each device participants receive.
Determine if adjunctive ERT treatment improves overall emotional distress greater than LVR alone measured by the Generalized Anxiety Disorder (GAD)-7 | 6 months
  The 7-item GAD-7 will measure symptoms of anxiety. Items are scored not at all (0) -Nearly every day (3), scores range from 0-21. Higher scores indicate more symptoms of anxiety.
Determine if adjunctive ERT treatment improves overall emotional distress greater than LVR alone measured by the Rumination-Reflection Questionnaire (RRQ) | 6 months
  The Rumination-Reflection Questionnaire is a 24-item measure of self-reflection tendencies. Items are scored from strongly disagree (1) - Strongly agree (5). Scores range from 24 to 120; a higher score means a worse outcome.
Determine if adjunctive ERT treatment improves overall emotional distress greater than LVR alone measured by the Penn State Worry Questionnaire (PSWQ) | 6 months
  The Penn State Worry Questionnaire is a 16-item self-report scale designed to measure the trait of worry in adults. Items are scored from not at all typical of me (1) - Very typical of me (5). The range of scores are from 16-80 with higher scores indicating higher level of worry.

CONTACTS AND LOCATIONS:
Overall Officials: K. Thiran Jayasundera, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No